CLINICAL TRIAL: NCT04610632
Title: Home Pregnancy Test Study Lay User Study on BioBank Samples
Brief Title: Home Pregnancy Test Study on BioBank Samples
Status: Completed | Type: Observational
Sponsor: SPD Development Company Limited (Industry)
Responsible Party: Sponsor
Other Study IDs: PROTOCOL-1147
Record Dates: First submitted 2020-10-27; First posted 2020-10-30 (Actual); Last update posted 2020-11-13 (Actual); Status verified 2020-11

CONDITIONS: Pregnancy Related

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: home pregnancy test — use of home pregnancy test

SUMMARY:
This is a non-clinical lay user study using stored clinical samples from the SPD BioBank.

Volunteers recruited into the study and meeting the criteria will test a randomised pregnant or not pregnant urine sample sourced from SPD's biobank with a new home pregnancy test. Volunteers will be required to follow the product instructions for use (IFU).

The order of testing will be randomised prior to execution of the protocol, and each urine sample will only be identifiable by a unique reference number. An independent study technician not involved in study conduct will be responsible for blinding the samples.

DETAILED DESCRIPTION:
Women will be informed of the opportunity to participate in a study in which they will be required to use a home pregnancy test to test a urine sample provided to them. Interested applicants will be invited to join the study.

Volunteers will be advised that the product they will be testing is under investigation and that the volunteer will not be testing their own urine and therefore volunteers will not learn their own pregnancy status.

Volunteers will be required to consent to the study prior to participation. Each volunteer will test only one device, they will be provided with one investigational device and one urine sample. The order of testing will be randomised prior to execution of the protocol, and each urine sample will only be identifiable by a unique reference number.

When ready the volunteer will be required to read the IFU prior to testing the urine sample provided with the investigational device according to the instructions. The volunteer will advise the study technician of the result, who will record this on the result sheet.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Aged ≥18 years
* Willing to give informed consent

Exclusion Criteria:

* Currently or previously employed by SPD, Abbott, Alere, Unipath, P&G or affiliates
* Has an immediate relative currently or previously (within last 5 years) employed by SPD, Abbott, Alere, Unipath or P&G or affiliates
* Is a qualified or trainee Healthcare Professional (HCP)
* Has professional experience of using dipstick type tests or lateral flow devices
* Has previously taken part in this study
* Seen the product within the past 6 months

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: General public
Sampling Method: Probability Sample
Enrollment: 81 (Actual)
Dates: Start 2020-11-09 (Actual); Primary Completion 2020-11-11 (Actual); Study Completion 2020-11-11 (Actual)

PRIMARY OUTCOMES:
Agreement with confirmed pregnancy result | 1 week
  The percentage agreement between the result obtained when a lay user test a urine sample, and the confirmed pregnancy status of the volunteer providing the sample. Both confirmed positive (pregnant) and negative (not pregnant) samples will be included in the study.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Johnson, Study Director — SPD Development Company Ltd
Locations (1):
- SPD Development Company Ltd., Bedford, Bedfordshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No